CLINICAL TRIAL: NCT04837898
Title: The Influence of Haskap Berry on Exercise Performance
Brief Title: Haskap and Endurance Running Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Mibelle Group Biochemistry (Industry); Haskapa Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26514
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2021-04

CONDITIONS: Exercise Performance
Keywords: berry; running; time trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplement will be pre-weighed by an individual (independent of the study) and provided to participants in sealed packets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haskap berry (Active Comparator): A commercially available haskap berry freeze-dried) powder
  Interventions: Dietary Supplement: Haskapa
- Placebo (Placebo Comparator): Black cherry KoolAid (Kraft Foods, USA) with added maltodextrin to match carbohydrate and calorie content
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Haskapa — Haskapa Ltd, Oxford, UK
  Arms: Haskap berry
Dietary Supplement: Placebo — isocaloric to the haskap powder
  Arms: Placebo

SUMMARY:
This study will employ a randomised, double-blind, placebo-controlled, independent groups experimental design. Submaximal, maximal and 5 km time trial running performance will be assessed before and after supplementation with haskap berry or a placebo.

DETAILED DESCRIPTION:
Participants will consume haskap berry powder or an isocaloric placebo for 7 days. They will be required to run on a treadmill before and after supplementation to asses the influence on the intervention on aerobic performance parameters. Other performance parameters such as blood lactate, heart rate, ratings of perceived exertion and respiratory variables will also be monitored throughout the various elements of the exercise trials.

ELIGIBILITY:
Inclusion Criteria:

* healthy non-smoking males
* completed a 5 km run (in less than 25 minutes) within the 6 weeks prior to the study

Exclusion Criteria:

* female
* allergies to fruit or dairy, currently taking any nutritional supplements (e.g. vitamins, antioxidant, herbal or sports enhancing supplements) or medication that might affect the study outcome
* history of gastrointestinal, renal or cardiovascular disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
5km time trial | Change from baseline at 7 days
  time to complete the trial (seconds)
V̇O2peak test | Change from baseline at 7 days
  time to exhaustion (seconds)

SECONDARY OUTCOMES:
Blood lactate response during submaximal tests, maximal and time trial | Change from baseline at 7 days
  lactate (mmol/L)
rating of perceived exertion during submaximal tests, maximal and time trial | Change from baseline at 7 days
  RPE (/20)
heart rate during submaximal tests, maximal and time trial | Change from baseline at 7 days
  (BPM)
VO2 during submaximal tests, maximal tests | Change from baseline at 7 days
  (oxygen uptake - relative ml/kg/min and absolute l/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be held by on a secure data based by the PI and made available to others but in line with contractual agreements with the funder and legal requirements of General Data Protection Regulations (GDPR) in the UK.